CLINICAL TRIAL: NCT06861543
Title: A Single Arm, Open Label, Dose-escalating, Prospective Phase I Clinical Trial Evaluating the Safety, Tolerability and Efficacy of TMT101 Injection Alone in Patients With Advanced Pancreatic Cancer or Non-small Cell Lung Cancer(NSCLC) After Standard Treatment Failure
Brief Title: The Purpose of This Study is to Evaluate the Safety, Tolerability and Efficacy of TMT101 Injection Monotherapy in Patients With Advanced Pancreatic Cancer or Non-small Cell Lung Cancer(NSCLC)
Acronym: TMT101-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wu Wenming, Director, Chief Physician of Basic Surgery, Principal Investigator, Clinical Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMT101-01
Record Dates: First submitted 2025-02-08; First posted 2025-03-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: TMT101 Injection; mRNA; advanced pancreatic cancer or NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: TMT101 Injection alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMT101 Injection monotherapy (Experimental): Three dose levels are planned to be explored: 0.1 mg, 0.2 mg, and 0.4 mg. The initial dose is 0.1 mg with a dose reduction for safety reasons, the level of dose reduction will be discussed jointly between the investigator and the sponsor. TMT101 will be injected intramuscularly, Once a week,a total of 9 times
  Interventions: Biological: TMT101 Injection

INTERVENTIONS:
Biological: TMT101 Injection — Three dose levels are planned to be explored: 0.1 mg, 0.2 mg, and 0.4 mg. The initial dose is 0.1 mg with a dose reduction for safety reasons, the level of dose reduction will be discussed jointly between the investigator and the sponsor. TMT101 will be injected intramuscularly, Once a week,a total of 9 times

SUMMARY:
This is a first-in-human, single-arm, open-label, dose escalation prospective phase I clinical study to evaluate the Safety, Tolerability and Efficacy of TMT101 Injection Alone in patients with Unresectable, Metastatic or Advanced pancreatic cancer or Non-small Cell Lung Cancer(NSCLC) after Standard Treatment Failure. The primary objective is to evaluate the safety and tolerability of TMT101 Injection as monotherapy in patients with advanced pancreatic cancer and NSCLC, and to determine the recommended therapeutic dose (RD) of TMT101 Injection as monotherapy

DETAILED DESCRIPTION:
The dose escalation trial adopts the "3+3" design , and about 3~6 patients with advanced pancreatic cancer or non-small cell lung cancer are enrolled in each dose level to evaluate the safety of TMT101 Injection alone. Three dose levels are planned to be explored: 0.1 mg, 0.2 mg, and 0.4 mg. Once a week, intramuscular Injection , a total of 9 times (the first tumor assessment is performed in the 6th week (±7 days), the investigator can decide the follow-up medication arrangement according to the tumor evaluation results). Dose-limiting toxicities (DLTs) will be assessed for each dose level, and the DLT observation period will be within 21 days from the first dose. The initial dose is 0.1 mg with a dose reduction for safety reasons, the level of dose reduction will be discussed jointly between the investigator and the sponsor. If the highest dose level of 0.4 mg is not confirmed as a possible recommended therapeutic dose (RD), it may be escalated a higher dose to determine the possible RD under the condition that investigator and the sponsor to decide together

ELIGIBILITY:
Inclusion Criteria:

1. Agrees to follow the trial protocol and visit schedule, has signed informed consent;
2. Subjects must be ≥18 years of age at time of informed consent,regardless of gender;
3. Patients with advanced/unresectable or metastatic pancreatic cancer or non-small cell lung cancer that requires histologically and/or cytologically confirmed according to the American Joint Committee on Cancer 8th edition; pancreatic cancer:Previous failure or intolerance of two or more lines of chemotherapy; NSCLC:Previous failure or intolerance of platinum-containing chemotherapy and anti-PD-1/PD-L1 monoclonal antibodies, regardless of combination therapy or sequential therapy, if the previous test for EGFR-sensitive mutations or ALK fusion genes is positive, treatment with a third-generation TKI must be failed or intolerant;
4. At least one evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
5. ECOG≤1;
6. Estimated life expectancy≥12 weeks;
7. Adequate organ function, meet the following laboratory standards:

   1. ANC≥1.5×109/L;PLT≥90×109/L;
   2. Hb≥90 g/L;
   3. TBIL≤1.5×ULN, Patients with Gilbert's syndrome ; without liver metastases, AST and ALT ≤ 2.5×ULN;liver metastases, AST and ALT ≤5×ULN ;
   4. Ccr≥50 mL/min;
   5. INR≤1.5×ULN, APTT≤1.5×ULN;
8. Males of childbearing potential and females of childbearing potential who are willing to use effective contraception since signing the informed consent until 6 months after the last dose of the trial drug. Females of childbearing potential must have a negative pregnancy test result within 7 days prior to the first dose.

Exclusion Criteria:

1. Allergic to TMT101 Injection or any of the components in the prescription;
2. Uncontrolled illness including, but not limited to, active infection requiring systemic therapy, uncontrolled hypertensionuncontrolled hyperglycemia, decompensated congestive heart failure , unstable angina, arrhythmias that require clinical intervention; ascites or uncontrolled pleural effusion (CTCAE 5.0≥grade 2), thrombosis (such as pulmonary embolism, cerebral infarction, myocardial infarction) or history of stroke, active autoimmune disease, psychiatric disease, active peptic ulcer disease, active bleeding disorder, which would limit compliance with study requirements or impair the patient's ability to sign informed consent in writing;
3. Patients who used immunosuppressive drugs within 3 weeks prior to the first dose, or patients who have achieved immunosuppressive intent (dose > 10 mg/day prednisone or other equivalent hormones and the duration of use is at least 7 days ) on systemic hormonal therapy or absorbable topical hormonal therapy, with the exception of physiologic doses of intranasal and inhaled corticosteroids;
4. Within 4 weeks prior to the first administration, received major surgery, radiotherapy (except palliative radiotherapy for bone metastasis), or treatment for surgical wounds that were not healed, ulcerated, or fractured; within 4 weeks prior to the first administration or within 5 half-lives (whichever is shorter) received anti-tumor treatments such as chemotherapy, biological therapy, endocrine therapy, targeted therapy, or immunotherapy.
5. Patients with prior or concurrent occurrence of other malignancies, with the following exceptions: a) Carcinoma in situ of the cervix or breast, curatively treated with no signs of recurrence for at least 3 years prior to the study; b) The primary malignancy was completely resected and in complete remission for ≥ 5 years;
6. History of interstitial lung disease or current interstitial lung disease or suspected of such disease by imaging during screening. and pneumonitis that previously required systemic corticosteroid treatment;
7. Treponema pallidum antibody or human immunodeficiency virus (HIV) antibody positive, positive for hepatitis C virus antibody and hepatitis C virus (HCV) RNA, or active hepatitis B (positive for hepatitis B surface antigen and HBV DNA ≥ upper limit of normal);
8. Received live vaccines within 4 weeks before the first dose or planned to receive live vaccines during the study period and within 4 weeks after the last dose, including but not limited to: measles, mumps, rubella, chickenpox, yellow fever, rabies, BCG and typhoid vaccines;
9. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
10. Interventional therapy in other clinical trials 3 weeks before the first dose, and it is judged by the investigator and medical monitor to be unsuitable for inclusion in the study;
11. Patients who have had a previous ≥grade 3 immune-related adverse event or immunotherapy-related serious adverse event (SAE) leading to permanent discontinuation;
12. Pregnant or lactating females;
13. In the opinion of the investigator, the subject has other conditions that may affect compliance or are not suitable for participation in this study;
14. Patient has active central nervous system metastases (with or without treatment), including symptomatic brain metastases or meningeal metastases or spinal cord compression, but asymptomatic brain metastases except;
15. Within 4 weeks prior to the first dose, all toxicities from prior antineoplastic therapy have not recovered to grade 1 or less, with the following exceptions: a. alopecia, b. long-term toxicity caused by radiotherapy, c. other toxicities that cannot be recovered in the judgment of the investigator but have no effect on the subject's administration
16. Major surgery within 4 weeks prior to the first dose;
17. Transsplenectomy which is not suitable is judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — regardless of gender
Enrollment: 18 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicities (DLTs) | within 21 days since the first dose
  Occurrence of dose-limiting toxicities (DLTs) within 21 days since the first dose
treatment-emergent adverse events (TEAEs) | up to 2 years
  occurrence of treatment-emergent adverse events (TEAEs) and grade according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
treatment related adverse event (TRAE) | up to 2 years
  Occurrence and grade of treatment related adverse event (TRAE) according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
immune-related Adverse Event(irAE） | up to 2 years
  Occurrence and grade of immune-related Adverse Event(irAE）according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Serious Adverse Event(SAE） | up to 2 years
  Occurrence and grade of Serious Adverse Event(SAE）according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Recommended Dose（RD） | the whole escalation phase within 21 days since the first dose
  During the dose escalation phase, the MTD and/or available safety, biomarker, and efficacy data will be evaluated thoroughly to determine the RD of TMT101 Injection alone . Three dose levels are planned to be explored: 0.1 mg, 0.2 mg, and 0.4 mg. Once the initial dose is 0.1 mg with a dose reduction for safety reasons, the level of dose reduction will be discussed jointly between the investigator and the sponsor. If the highest dose level of 0.4 mg is not confirmed as a possible recommended therapeutic dose (RD), it may be escalated to a higher dose to determine the possible RD under the condition that investigator and the sponsor to decide together.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and iRECIST
Disease control rate (DCR) | up to 2 years
  the percentage of patients with CR or PR or stable disease (SD) as BOR according to RECIST v1.1 and iRECIST divided by the number of patients in the efficacy analysis set
Progression-free survival (PFS) | up to 2 years
  the time of first trial treatment until the first objective tumor progression according to RECIST v1.1 and iRECIST or death from any cause, whichever occurs first
Overall survival (OS) | up to 2 years
  the time of first trial treatment until death from any cause
Peak time (Tmax) of cationic lipids | up to 9 weeks
Peak concentration (Cmax) of cationic lipids | up to 9 weeks
Area under the drug concentration -time curve (AUC) of cationic lipids | up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Wu, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China